CLINICAL TRIAL: NCT05607537
Title: An Open-Label, Single-Center, 2-Part, Parallel Study to Determine the Absolute Bioavailability and the Absorption, Metabolism, and Elimination Properties of [14C]E7386 in Healthy Male Subjects
Brief Title: A Study to Determine the Absolute Bioavailability and the Absorption, Metabolism, and Elimination Properties of Carbon-14 (14C)E7386 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E7386-E044-003; 2022-000954-27 (EudraCT Number)
Record Dates: First submitted 2022-10-14; First posted 2022-11-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers
Keywords: E7386
MeSH Terms: interventions — E-7386

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: E7386 40 mg Tablet + (14C)E7386 (Experimental): Participants will be administered a single oral dose of E7386 40 mg tablet on Day 1 followed by an intravenous infusion containing a microdose solution of [14C]E7386 (100 mcg) with not more than (NMT) 7.4 kilobecquerel (kBq) (0.20 microcurie [mcCi]), starting approximately 25 minutes post oral dose administered as 5 milliliter (mL) over 5 minutes to coincide with the time at which the highest drug concentration occurs (tmax) for E7386 after an oral dose.
  Interventions: Drug: E7386 Tablet; Drug: (14C)E7386
- Part 2: (14C)E7386 40 mg Capsule (Experimental): Participants will be administered a single oral dose of E7386 40 mg capsule radiolabeled with approximately 2.96 megabecquerel (MBq) (80 mcCi) (14C)E7386 (final dose to depend on the specific activity of [14C]E7386) in the morning on Day 1 after an overnight fasting.
  Interventions: Drug: (14C)E7386 Capsule

INTERVENTIONS:
Drug: E7386 Tablet — E7386 40 mg tablet.
  Arms: Part 1: E7386 40 mg Tablet + (14C)E7386
Drug: (14C)E7386 Capsule — (14C)E7386 40 mg capsule.
  Arms: Part 2: (14C)E7386 40 mg Capsule
Drug: (14C)E7386 — (14C)E7386 administered intravenously.
  Arms: Part 1: E7386 40 mg Tablet + (14C)E7386

SUMMARY:
The primary purpose of this study is to evaluate the absolute bioavailability of E7386 following a single oral dose of E7386 as a one 40 milligram (mg) immediate release (IR) tablet and concomitant intravenous (IV) microdose of (14C)E7386 (100 mcg [microgram]) solution for Part 1 and to determine the pharmacokinetic (PK) and excretion of E7386 following a single 40 mg powder in capsule (PIC) oral administration of (14C)E7386 for Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, healthy male, age greater than or equal to (>=) 30 years and less than or equal to (<=) 55 years old at the time of informed consent
2. Body Mass Index (BMI) of greater than (>) 18 to less than (<) 30 kilogram per square meter (kg/m^2) as measured at Screening
3. Adequate organ function per blood work
4. Participant must have regular bowel movements (that is, average stool production of >=1 and <=3 stools per day)
5. Participant must agree to adhere to the contraception requirements

Exclusion Criteria:

1. Have participated in any clinical research study involving nonradiolabeled investigational product within 90 days prior to Day -1 (Baseline) or involving radiolabeled investigational product within 12 months prior to Day -1 (Baseline)
2. Participant has had exposure to significant diagnostic or therapeutic radiation (example, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to Day -1 (Baseline)
3. Male participant with pregnant or breastfeeding partner
4. Male participant who is unwilling to follow the contraception rules of the study for up to 92 days after last dose of the study drug
5. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks prior to dosing
6. A prolonged QT/QTc interval (QTcF [corrected QT interval by Fridericia] >450 millisecond [ms]) as confirmed by a repeated ECG at Screening or Baseline, or a history of risk factors for torsade de pointes (example, heart failure, hypokalemia, family history of long QT Syndrome), or the use of concomitant medications that prolonged the QT/QTc interval
7. Known history of clinically significant drug, food allergies, or presently experiencing any seasonal or perennial allergy at Screening and Baseline (Day -1)
8. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb) or human immunodeficiency virus (HIV) antibody at Screening
9. History of recreational drug use, drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive urine drug test or breath alcohol test at Screening or admission
10. Participant who is, or is an immediate family member of, a study site or sponsor employee
11. Participant does not have suitable veins for multiple venipunctures/cannulations as assessed by the investigator or delegate at Screening
12. Receipt of blood products within 4 weeks prior to dosing, or donation of blood or plasma within the previous 3 months, or loss of greater than 400 mL of blood
13. Any history of or concomitant medical condition that in the opinion of the investigator would compromise the participant's ability to safely complete the study at Screening and Day -1 (Baseline)
14. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Part 1, %F: Percent Absolute Oral Bioavailability for (14C)E7386 and E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, Cmax: Maximum Observed Plasma Concentration for Total Radioactivity, (14C)E7386 and E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, Tlag: Time Delay Between Drug Administration and the Onset of Absorption for Total Radioactivity, (14C)E7386 and E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, Tmax: Time to Reach Maximum Observed Plasma Concentration (Cmax) for Total Radioactivity, (14C)E7386 and E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, AUC(0-12h): Area Under the Plasma Concentration-time Curve From Time Zero to 12 hours Post-dose for Total Radioactivity, (14C)E7386 and E7386 | Pre-dose (0 hour) up to 12 hours post-dose
Part 1, AUC(0-24h): Area Under the Plasma Concentration-time Curve From Time Zero to 24 hours Post-dose for Total Radioactivity, (14C)E7386 and E7386 | Pre-dose (0 hour) up to 24 hours post-dose
Part 1, AUC(0-last): Area Under the Plasma Concentration-time Curve from Time 0 to Time of the Last Measurable Concentration for Total Radioactivity, (14C)E7386 and E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time Zero to Infinite Time for Total Radioactivity, (14C)E7386 and E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, t1/2: Apparent Terminal Elimination Phase Half-life for Total Radioactivity, (14C)E7386 and E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, MRT: Mean Residence Time of (14C)E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, CL: Total Clearance of (14C)E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, CL/F: Apparent Total Body Clearance of E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, Vss: Volume of Distribution at Steady State of (14C)E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, Vz/F: Apparent Volume of Distribution at Terminal Phase of E7386 | Pre-dose (0 hour) up to 96 hours post-dose
Part 1, Fa: Percentage of Absorbed Dose Using Total Radioactivity in Urine | Pre-dose (0 hour) up to 96 hours post-dose
Part 2, Cmax: Maximum Observed Concentration for Total Radioactivity and E7386 | Pre-dose (0 hour) up to 480 hours post-dose
Part 2, Tlag: Time Delay Between Drug Administration and the Onset of Absorption for Total Radioactivity and E7386 | Pre-dose (0 hour) up to 480 hours post-dose
Part 2, Tmax: Time to Reach Maximum Observed Concentration (Cmax) for Total Radioactivity and E7386 | Pre-dose (0 hour) up to 480 hours post-dose
Part 2, AUC(0-12h): Area Under the Concentration-time Curve From Time Zero to 12 hours Post-dose for Total Radioactivity and E7386 | Pre-dose (0 hour) up to 12 hours post-dose
Part 2, AUC(0-24h): Area Under the Concentration-time Curve From Time Zero to 24 hours Post-dose for Total Radioactivity and E7386 | Pre-dose (0 hour) up to 24 hours post-dose
Part 2, AUC(0-last): Area Under the Concentration-time Curve from Time 0 to Time of the Last Measurable Concentration for Total Radioactivity and E7386 | Pre-dose (0 hour) up to 480 hours post-dose
Part 2, AUC(0-inf): Area Under the Concentration-time Curve From Time Zero to Infinite Time for Total Radioactivity and E7386 | Pre-dose (0 hour) up to 480 hours post-dose
Part 2, t1/2: Apparent Terminal Elimination Phase Half-life for Total Radioactivity and E7386 | Pre-dose (0 hour) up to 480 hours post-dose
Part 2, CL/F: Apparent Total Body Clearance of E7386 | Pre-dose (0 hour) up to 480 hours post-dose
Part 2, Vz/F: Apparent Volume of Distribution at Terminal Phase of E7386 | Pre-dose (0 hour) up to 480 hours post-dose
Part 2, feu: Percentage of Administered Radioactive Dose Excreted in Urine for Total Radioactivity | Day -1 (Baseline) up to Day 49
Part 2, Cumulative feu(0-tlast): Cumulative Radioactive Dose Excreted in Urine From Time 0 to Time of the Last Measurable Concentration | Day -1 (Baseline) up to Day 49
Part 2, fef: Percentage of Total Radioactivity Recovered in Feces Relative to the Administered Radioactive Dose | Day -1 (Baseline) up to Day 49
Part 2, Cumulative fef(0-tlast): Cumulative Radioactive Dose Excreted in Feces From Time 0 to Time of the Last Measurable Concentration | Day -1 (Baseline) up to Day 49
Part 2, feu+ef: Percentage of Total Radioactivity Recovered in Combined Urine and Feces Relative to the Administered Radioactive Dose | Day -1 (Baseline) up to Day 49
Part 2, Cumulative feu+ef(0-tlast): Cumulative Radioactive Dose excreted in Combined Excreta (Urine and Feces) From Time Zero to Time of the Last Measurable Concentration | Day -1 (Baseline) up to Day 49
Part 2, Fa: Percentage of Absorbed Dose Using Total Radioactivity in Urine | Day -1 (Baseline) up to Day 49

SECONDARY OUTCOMES:
Part 2 (Metabolic Profile of E7386): Concentration of Metabolite of E7386 in Plasma, Urine, and Feces | Day 1 up to Day 21
  Blood, urine and feces samples will be collected and analyzed to estimate the concentration of metabolite of E7386 by liquid chromatography/multiple-stage mass spectroscopy method.
Parts 1 and 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Part 1: Up to Day 5; Part 2: Up to Day 49
Parts 1 and 2: Number of Participants With Abnormal Laboratory Values | Part 1: Up to Day 5; Part 2: Up to Day 49
  Laboratory assessment will include hematology, clinical chemistry, and urinalysis parameters.
Parts 1 and 2: Number of Participants With Abnormal Vital Signs Values | Part 1: Up to Day 5; Part 2: Up to Day 49
  Vital sign measurements will include systolic and diastolic blood pressure (BP), pulse rate, respiratory rate, body temperature.
Parts 1 and 2: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Values | Part 1: Up to Day 5; Part 2: Up to Day 49
Parts 1 and 2: Number of Participants With Abnormal Ophthalmic Examinations | Part 1: Up to Day 5; Part 2: Up to Day 49
Parts 1 and 2: Number of Participants who will Receive Concomitant Medications | Part 1: Up to Day 5; Part 2: Up to Day 49
Parts 1 and 2: Number of Participants With Abnormal Physical Examinations | Part 1: Up to Day 5; Part 2: Up to Day 49
Parts 1 and 2: Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-suicide Severity Rating Scale (C-SSRS) | Part 1: Up to Day 5; Part 2: Up to Day 49
  The C-SSRS is an interview-based rating scale to systematically assess any suicidality, suicidal behavior, or suicidal ideation. Any suicidality is emergence of any suicidal ideation or suicidal behavior. Any suicidal behavior is indicated when response is "yes" for any these questions- actual attempt to suicide, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation is indicated when response is "yes" for any of these questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide.

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Clinical Research Unit, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.